CLINICAL TRIAL: NCT00203645
Title: Minimal and Brief Treatments for Pathological Gamblers: Developing Effective Treatment Systems
Brief Title: Minimal and Brief Treatments for Pathological Gamblers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: David Hodgins, UCalgary
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 110328 - CIHR; 1016 - OPGRC
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Pathological Gambling
Keywords: Problem gambling; Self-help manual; Motivation enhancement; Telephone support; Treatment; Pathological gambling
MeSH Terms: conditions — Gambling | interventions — Bibliotherapy; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Brief self-directed treatment (Experimental): self-help workbook plus motivational telephone intervention
  Interventions: Behavioral: Self-help treatment
- Self-directed plus telephone support (Experimental): Self-help workbook, motivational telephone intervention plus telephone booster calls
  Interventions: Behavioral: Self-help treatment
- Workbook only (Active Comparator): Workbook only
  Interventions: Behavioral: Self-help treatment
- Waitlist (No Intervention): Six week waitlist

INTERVENTIONS:
Behavioral: Self-help treatment — Workbook "Becoming a Winner",
  Other Names: Bibliotherapy; motivational interviewing
  Arms: Brief self-directed treatment; Self-directed plus telephone support; Workbook only

SUMMARY:
The purpose of the study is to examine whether problem gamblers who receive therapy calls in addition to a self-help manual will be more likely to quit or cut back on their gambling when compared with problem gamblers who receive just the manual.

DETAILED DESCRIPTION:
With gambling becoming more accessible, the occurrence of problems related to gambling are on the rise. The costs of problem gambling are enormous.There are social and economic costs, the gambler can sometimes lose a significant relationship, job, or commit an illegal activity. Pathological gamblers are also at risk for developing a general medical condition related to stress. There is a high risk of suicide and problem gamblers also have increased rates of mental health disorders. Relatively few people choose to attend formal treatment programs so it's important to provide a range of options to make treatment more accessible. The present study examines the effectiveness of minimal and brief interventions delivered by the telephone.

Comparison(s): The "Workbook Only Control" condition involves receiving the self-help booklet through the mail after a brief telephone assessment. The "Minimal Treatment" condition involves receiving the same workbook but also having a motivational enhancement intervention by telephone. The "Brief Treatment" condition provides the workbook, motivational enhancement, and follow-up support on six occasions spread over 36 weeks. The "Wait List Control" condition involves participants being assigned to a six week waiting list. Participants are assessed and after a six week waiting period they will have a reassessment at which time they will be sent the gambling self-help workbook.

ELIGIBILITY:
Inclusion Criteria:

* Over age 17
* Perception of a gambling problem and a score of 3 or higher (moderate risk) on the Canadian Problem Gambling Index.
* Not involved in treatment at present.
* Willingness to read a short book written in English as a major treatment.
* Willing to have telephone contacts recorded.
* Willing to provide follow-up data on gambling.
* Willing to provide the name of a collateral to help locate them for follow-up interviews.
* Must have gambled at least once in the past month

Exclusion Criteria:

* Participants in the preliminary study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2003-07; Primary Completion 2006-04 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Days of Gambling | 3,6,9 12 months
Money lost | 3,6,9 12 months

SECONDARY OUTCOMES:
Gambling problem severity | 12 months
Psychiatric symptoms | 12 months
Self-efficacy | 3,6,9,12 months

CONTACTS AND LOCATIONS:
Overall Officials: David C Hodgins, PhD., Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Hodgins DC, Currie SR, el-Guebaly N. Motivational enhancement and self-help treatments for problem gambling. J Consult Clin Psychol. 2001 Feb;69(1):50-7. doi: 10.1037//0022-006x.69.1.50. PMID 11302277
- [Background] Hodgins DC, Currie S, el-Guebaly N, Peden N. Brief motivational treatment for problem gambling: a 24-month follow-up. Psychol Addict Behav. 2004 Sep;18(3):293-6. doi: 10.1037/0893-164X.18.3.293. PMID 15482086